CLINICAL TRIAL: NCT04115358
Title: Clinical and Radiographic Evaluation of Formocresol, Ferric Sulfate and Hyaluronic Acid Pulpotomies on Human Primary Teeth: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Hyaluronic Acid Pulpotomies in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MarmaraPD
Record Dates: First submitted 2019-09-09; First posted 2019-10-04 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-02

CONDITIONS: Pulpitis
Keywords: Pulpotomy
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic acid (Experimental): Gengigel teething (%0,54 hyaluronic acid), 0,1ml to the orifice of the root canals of the primary molar.
  Interventions: Procedure: Hyaluronic acid: Gengigel teething
- Formocresol (Active Comparator): 0,1 ml to the orifice of the root canals of the primary molar.
  Interventions: Procedure: Formocresol Buckley formula: Formacresol
- Ferric sulfate (Active Comparator): 0,1 ml to the orifice of the root canals of the primary molar.
  Interventions: Procedure: Ferric sulfate: ViscoStat

INTERVENTIONS:
Procedure: Hyaluronic acid: Gengigel teething — Applying of 0,54% hyaluronic acid for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns and composite filling material.
  Arms: Hyaluronic acid
Procedure: Formocresol Buckley formula: Formacresol — Applying of 1/5 diluted formocresol for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns and composite filling material.
  Arms: Formocresol
Procedure: Ferric sulfate: ViscoStat — Applying of 20% ferric sulfate for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns and composite filling material.
  Arms: Ferric sulfate

SUMMARY:
In this study, 120 primary molar teeth from healthy children aged between 5 and 9 and who apply to Marmara University Faculty of Dentistry, Department of Pediatric Dentistry will be subjected to pulpotomy treatments. After proper diagnosis of coronal pulpitis, the teeth will be assigned randomly to one of the 3 groups: 40 primary molars for formocresol (FC) pulpotomy treatments, 40 primary molars for ferric sulfate (FS) treatments and 40 primary molars for 0.5% hyaluronic acid gel (HA) pulpotomy treatments. The tooth decay will be removed, the pulp will be amputated from the chamber of the pulp with a sharp excavator and one of the medicament will be applied to the orifice of the root canals. The cavity will be sealed tight with zinc oxide cement, and the primary molars will be restored with a composite filling material or with a stainless steel crown (SSC). A single investigator will perform the procedure. The teeth will be followed clinically and radiographically at 1st, 3rd, 6th, 12th months.

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of the materials used in pulpotomies, and to evaluate the success of hyaluronic gel over the formocresol and/or ferric sulfate considered as the gold standard for this type of treatment.

Pulpotomy is an endodontic treatment method aiming to maintain primary molar affected from deep caries and acute pulpitis by removing the effected pulpal tissue, leaving the remaining root canal pulp and maintaining its vitality and function until the tooth exfoliates physiologically. In order to remain canals intact and uninflamed various dental materials are used according to treatment purposes; categorized into three groups as devitalizing, preventive and regenerative treatment.

1. Devitalization: Formocresol, Glutaraldehyde, Electro-surgery
2. Protective: Ferric Sulfate, Calcium Hydroxide, Mineral Trioxide Aggregate, Lasers
3. Regenerative: Bone Morphogenetic Protein, Enriched Collagen

The ideal agent or method for pulpotomy treatment of the primary teeth has not been determined yet but the earliest method of diluted formocresol is considered by many the gold standard. Formocresol is a strong strain that fixes living tissues. It contains formaldehyde gas, organic structures, dentin channels and narrow side channels until the bacteria are also fixed. 10% formalin solution (14% formaldehyde) is used as a tissue fixative.

Ferric Sulfate an other material for pulpotomy is used in dentistry mainly as a hemostatic agent. It has several advantages over formocresol such as non-mutagenic property and keeping root canal pulp vital.

Hyaluronic acid gel, which is a new product as a pulpotomy material, has been used in dentistry as well as medicine for many years. It is distributed widely in epithelial and connective tissues. Medical uses include joint treatments, skin lotions for atopic dermatitis, cosmetic surgery etc. In dentistry, gingivitis, teething, dental surgery including implants and sinus lifting procedures and oral ulcers are main target for hyaluronic acid treatment. This study extends the use of hyaluronic acid to primary tooth endodontics.

In this study, 120 primary molar teeth from healthy children aged between 5 and 9 and who apply to Marmara University Faculty of Dentistry Department of Pediatric Dentistry will be subjected to pulpotomy treatments. Sample size calculation showed that at first 40 teeth in each group will be required to detect a significant difference (80% power, two-sided 5% significance level).

Ethical approval of the study was taken from the Clinical Research Ethics Committee, Faculty of Dentistry at Marmara University (No: 2019/288) in accordance with the Declaration of Helsinki. The patients' family will be given information about the pros and cons of the study on the relevant teeth and then a written consent will be obtained.

Patients will be selected for this study according to the following criteria:

1. Children who have good cooperation, do not require general anesthesia or sedation, and who do not have any systemic disease, allergic reactions, or any use of medications.
2. No spontaneous, continuous pain in the tooth, no pathological or physiological mobility, no abscess and/or fistula, no tenderness to palpation or percussion.
3. The tooth can be restored with a stainless steel crown (SSC) or a composite filling material after treatment.
4. The physiological resorption in the tooth root not exceeding 1/3.
5. No pathological resorption in the tooth root canals internally and/or externally, no radiolucency in the periapical or furcation regions, no enlargement of periodontal ligaments.

Exclusion criteria:

1. Children who have any disorders, spontaneous pain, no restorable primary molars, may exfoliate soon and teeth with apical periodontitis, pulp necrosis, abscess, fistula, swelling or mobility.
2. Families who are not willing to join the study.

After proper diagnosis of coronal pulpitis, local anesthesia is administrated, the teeth will be assigned randomly to one of the 3 groups: 40 primary molars for formocresol pulpotomy treatments, 40 primary molars for ferric sulfate treatments and 40 primary molars for 0.5% hyaluronic acid gel pulpotomy treatments. The tooth decay is removed, the roof of the pulp chamber is removed by joining the pulp horns with a bur cut. The coronal pulp is amputated from the chamber of the pulp with a sharp excavator and one or more cotton pellets is placed over the site and pressure is applied. When the hemostasis is insured, one of the medicament is applied to the orifice of the root canals. The cavity will be sealed tight with zinc oxide eugenol cement. The primary molars were restored either with a stainless-steel crown in case of proximal cavities or with a composite filling material in case of occlusal cavities. A single pediatric dentist will perform whole pulpotomy treatments and restorations of all selected teeth. The teeth will be followed clinically and radiographically at 1, 3, 6, 12 months.

The teeth will be evaluated clinically and radiographically according to the following criteria:

1. Clinical criteria: Spontaneous pain, tenderness to percussion and/or palpation, pathological mobility and abscess or fistula.
2. Radiographic criteria: Periapical or furcal radiolucency, internal or external root resorption, loss of lamina dura.

All evaluations will be performed by two calibrated pediatric dentists. The performing dentist will not be blinded to the treatment materials but the patient and two examiners who evaluated clinical and radiographic findings will be blinded to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease,
* No pathological mobility and/or resorption of the tooth,
* No pain and/or abscess,
* Parents volunteering,
* The patients are between 5-9 years old.

Exclusion Criteria:

* Systemic disease,
* Pathological mobility and resorption of the tooth,
* Pain and/or abscess,
* Non voluntary,
* The patients aren't between 5-9 years old.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mentes, Prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Pediatric Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in May 2019 and the last participant was enrolled in September 2019. No important changes in methods or selection criteria have been done. 1st, 3rd and 6th months assessments were made without complications but 1-year examination had some face to face problems with the Covid-19 pandemics. So some final examinations and patient comforts had been done via phone and/or online connections.
Pre-assignment Details: The study was initially carried out on 136 primary molars of 47 children. Three children (2 boys, 1 girl) did not show up in any recalls, so the study was performed in 130 primary molars.
Units Other Than Participants: teeth
Groups:
- Hyaluronic Acid: Gengigel teething (%0,54 hyaluronic acid), 0,1ml to the orifice of the root canals of the primary molar
  Hyaluronic acid: Gengigel teething: Applying of 0,54% hyaluronic acid for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown and composite filling material.
- Formocresol: 0,1 ml to the orifice of the root canals of the primary molar.
  Formocresol Buckley formula: Formacresol: Applying of 1/5 diluted formocresol for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown and composite filling material.
- Ferric Sulfate: 0,1 ml to the orifice of the root canals of the primary molar.
  Ferric sulfate: ViscoStat: Applying of 20% ferric sulfate for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown and composite filling material.
Period: Overall Study
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Started | 34; 51 teeth | 33; 40 teeth | 34; 39 teeth
Completed (In the 12th month follow-up, the dropouts increased due to the Covid-19 pandemic and periapical radiographs could not be taken in a total of eight children.) | 34; 48 teeth (34 participants 48 teeth for clinical assessment, 28 participants 35 teeth for radiographic assessment.) | 33; 40 teeth (33 participants 40 teeth for clinical assessment, 26 participants 32 teeth for radiographic assessment.) | 33; 38 teeth (34 participants 38 teeth for clinical assessment, 26 participants 31 teeth for radiographic assessment.)
Not Completed | 0; 3 teeth | 0; 0 teeth | 1; 1 teeth
Not completed — exfoliation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: same participant can have more that 1 tooth (unit).
Units Other Than Participants: tooth
Groups:
- Hyaluronic Acid: Gengigel teething (%0,54 hyaluronic acid), 0,1ml to the orifice of the root canals of the primary molar.
  Hyaluronic acid: Gengigel teething: Applying of 0,54% hyaluronic acid for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns (SSC) and composite filling material.
- Formocresol: 0,1 ml to the orifice of the root canals of the primary molar
  Formocresol Buckley formula: Formacresol: Applying of 1/5 diluted formocresol for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns (SSC) and composite filling material.
- Ferric Sulfate: 0,1 ml to the orifice of the root canals of the primary molar
  Ferric sulfate: ViscoStat: Applying of 20% ferric sulfate for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crowns (SSC) and composite filling material.
- Total: Total of all reporting groups
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate | Total
Number analyzed (Participants) | 34 | 33 | 34 | 101
Number analyzed (tooth) | 51 | 40 | 39 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 33 | 34 | 101
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.65 (0.99) | 6.83 (0.98) | 6.67 (1.08) | 6.71 (1.015)
Sex: Female, Male [Count of Units; unit: tooth]
  Female | 32 | 25 | 23 | 80
  Male | 19 | 15 | 16 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    (all) |  |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 34 | 33 | 34 | 101
Dental Arch/Tooth Type [Count of Units; unit: tooth]
  Maxillary 1st primary molars | 11 | 9 | 7 | 27
  Maxillary 2nd primary molars | 17 | 13 | 8 | 38
  Mandibular 1st primary molars | 14 | 11 | 15 | 40
  Mandibular 2nd primary molars | 9 | 7 | 9 | 25
Dental Arch [Count of Units; unit: tooth]
  Lower Arch | 23 | 18 | 24 | 65
  Upper Arch | 28 | 22 | 15 | 65
Tooth Type [Count of Units; unit: tooth]
  1st primary molars | 25 | 20 | 22 | 67
  2nd primary molars | 26 | 20 | 17 | 63
Final Restoration [Count of Units; unit: tooth]
  SSC | 33 | 28 | 28 | 89
  Composite | 18 | 12 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Teeth Sensitive to Percussion in 3 Groups
Description: Sensitivity to biting, chewing and clinically to the percussion by a probe
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Groups:
- Hyaluronic Acid: Gengigel teething (%0,54 hyaluronic acid), 0,1ml to the orifice of the root canals of the primary molar
  Hyaluronic acid: Gengigel teething: Applying of 0,54% hyaluronic acid for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown or composite filling material.
- Formocresol: 0,1 ml to the orifice of the root canals of the primary molar
  Formocresol Buckley formula: Formacresol: Applying of 1/5 diluted formocresol for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown or composite filling material.
- Ferric Sulfate: 0,1 ml to the orifice of the root canals of the primary molar
  Ferric sulfate: ViscoStat: Applying of 20% ferric sulfate for one minute to the orifice of root canals of the primary molars, then sealing the chamber with zinc oxide eugenol cement and completing the restoration with stainless steel crown or composite filling material.
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 7 | 6 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

2. Primary Outcome: Number of Teeth Sensitive to Percussion in 3 Groups
Description: Sensitivity to biting, chewing and clinically to the percussion by a probe
Time Frame: Change from Baseline at 3 months in 3 groups
Population: 1 tooth is extracted in HA group so 50 teeth are evaluated
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 10 | 8 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

3. Primary Outcome: Number of Teeth Sensitive to Percussion in 3 Groups
Description: Sensitivity to biting, chewing and clinically to the percussion by a probe
Time Frame: Change from Baseline at 6 months in 3 groups
Population: 1 tooth exfoliated in FS group and 1 participant so no observation for 1 tooth and 1 participant in FS
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 11 | 8 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

4. Primary Outcome: Number of Teeth Sensitive to Percussion in 3 Groups
Description: Sensitivity to biting, chewing and clinically to the percussion by a probe
Time Frame: Change from Baseline at 12 months in 3 groups
Population: 2 teeth exfoliated from HA group (not participants) so number of teeth reduced from 50 to 48
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 48 | 40 | 38
teeth | 2 | 6 | 2
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

5. Primary Outcome: Number of Mobile Teeth in 3 Groups
Description: Mobility of the treated tooth and/or the tooth is sensitive to the vibration
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 1 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

6. Primary Outcome: Number of Mobile Teeth in 3 Groups
Description: Mobility of the treated tooth and/or the tooth is sensitive to the vibration
Time Frame: Change from Baseline at 3 month in 3 groups
Population: 1 tooth extracted from HA group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 1 | 0 | 1
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

7. Primary Outcome: Number of Mobile Teeth in 3 Groups
Description: Mobility of the treated tooth and/or the tooth is sensitive to the vibration
Time Frame: Change from Baseline at 6 month in 3 groups
Population: 1 tooth exfoliated from FS group (1 participant ) so 1 child and 1 tooth is reduced from FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 3 | 2 | 1
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

8. Primary Outcome: Number of Mobile Teeth in 3 Groups
Description: Mobility of the treated tooth and/or the tooth is sensitive to the vibration
Time Frame: Change from Baseline at 12 months in 3 groups
Population: 2 teeth exfoliated from HA group (not participants) so 50 teeth reduced to 48 teeth but participants still exist
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 48 | 40 | 38
teeth | 4 | 4 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

9. Primary Outcome: Number of Teeth With Patient Discomfort and/or Pain in 3 Groups
Description: Any pain history at that time frame and/or complaint of discomfort and pain clinically
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 1 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

10. Primary Outcome: Number of Teeth With Patient Discomfort and/or Pain in 3 Groups
Description: Any pain history at that time frame and/or complaint of discomfort and pain clinically
Time Frame: Change from Baseline at 3 months in 3 groups
Population: 1 tooth extracted from HA group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

11. Primary Outcome: Number of Teeth With Patient Discomfort and/or Pain in 3 Groups
Description: Any pain history at that time frame and/or complaint of discomfort and pain clinically
Time Frame: Change from Baseline at 6 months in 3 groups
Population: 1 tooth exfoliated (one participant) so 1 tooth and 1 participant are reduced from FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

12. Primary Outcome: Number of Teeth With Patient Discomfort and/or Pain in 3 Groups
Description: Any pain history at that time frame and/or complaint of discomfort and pain clinically
Time Frame: Change from Baseline at 12 months in 3 groups
Population: 2 teeth exfoliated in HA group so 50 teeth reduced to 48 but no participant is reduced
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 48 | 40 | 38
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

13. Primary Outcome: Number of Teeth With Dental Abscess in 3 Groups
Description: Any sign of chronic pulpitis, redness or swelling of the gingiva and/or fistula at that time frame and clinically
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 1 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

14. Primary Outcome: Number of Teeth With Dental Abscess in 3 Groups
Description: Any sign of chronic pulpitis, redness or swelling of the gingiva and/or fistula at that time frame and clinically
Time Frame: Change from Baseline at 3 months in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

15. Primary Outcome: Number of Teeth With Dental Abscess in 3 Groups
Description: Any sign of chronic pulpitis, redness or swelling of the gingiva and/or fistula at that time frame and clinically
Time Frame: Change from Baseline at 6 months in 3 groups
Population: 1 tooth exfoliated in FS group so 1 tooth and 1 participant are reduced in FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

16. Primary Outcome: Number of Teeth With Dental Abscess in 3 Groups
Description: Any sign of chronic pulpitis, redness or swelling of the gingiva and/or fistula at that time frame and clinically
Time Frame: Change from Baseline at 12 months
Population: 2 teeth exfoliated from HA group so number of teeth reduced from 50 to 48 but participants are same
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 48 | 40 | 38
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

17. Primary Outcome: Number of the Pathological Exfoliation of Affected Teeth in 3 Groups
Description: The tooth is missing or ready to exfoliate physiologically and no pathology is examined
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 0 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

18. Primary Outcome: Number of the Pathological Exfoliation of Affected Teeth in 3 Groups
Description: The tooth is missing or ready to exfoliate physiologically and no pathology is examined
Time Frame: Change from Baseline at 3 months in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 1 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

19. Primary Outcome: Number of the Pathological Exfoliation of Affected Teeth in 3 Groups
Description: The tooth is missing or ready to exfoliate physiologically and no pathology is examined
Time Frame: Change from Baseline at 6 months in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 0 | 0 | 1
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

20. Primary Outcome: Number of the Pathological Exfoliation of Affected Teeth in 3 Groups
Description: The tooth is missing or ready to exfoliate physiologically and no pathology is examined
Time Frame: Change from Baseline at 12 months in 3 groups
Population: 2 exfoliations in HA group are shown here
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 2 | 0 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

21. Primary Outcome: Number of Teeth With Root Resorption in 3 Groups
Description: Internal, external, early or physiological root resorption from periapical/panoramic radiographs
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth
  Periapical resorption | 1 | 1 | 2
  Internal resorption | 6 | 4 | 1
  External resorption | 1 | 0 | 1
  No resorption | 43 | 35 | 35
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

22. Primary Outcome: Number of Teeth With Root Resorption in 3 Groups
Description: Internal, external, early or physiological root resorption from periapical/panoramic radiographs
Time Frame: Change from Baseline at 3 months in 3 groups
Population: 1 tooth extracted in HA group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth
  Periapical resorption | 2 | 3 | 4
  Internal resorption | 9 | 11 | 6
  External resorption | 6 | 1 | 3
  No resorption | 33 | 25 | 26
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

23. Primary Outcome: Number of Teeth With Root Resorption in 3 Groups
Description: Internal, external, early or physiological root resorption from periapical/panoramic radiographs
Time Frame: Change from Baseline at 6 months
Population: 1 tooth exfoliated from FS group so 1 tooth and 1 participant reduced in FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth
  Periapical resorption | 7 | 5 | 5
  Internal resorption | 11 | 12 | 10
  External resorption | 5 | 5 | 5
  No resorption | 27 | 18 | 18
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

24. Primary Outcome: Number of Teeth With Root Resorption in 3 Groups
Description: Internal, external, early or physiological root resorption from periapical/panoramic radiographs
Time Frame: Change from Baseline at 12 months
Population: 6 participants, 12 teeth missing for xrays, 2 exfoliations from HA group; 7 participants, 8 teeth missing for xrays from FC group; 7 participants, 7 teeth missing for xrays from FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 28 | 26 | 26
Number analyzed (teeth) | 35 | 32 | 31
teeth
  Periapical resorption | 12 | 8 | 15
  Internal resorption | 11 | 8 | 5
  External resorption | 7 | 6 | 5
  No resorption | 5 | 10 | 6
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

25. Primary Outcome: Number of Teeth With Any Root Lesion From Radiography in 3 Groups
Description: Radiographic evaluation for any periapical or bifurcal lesion, cyst formation or obliteration
Time Frame: Change from Baseline at 1 month in 3 groups
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth | 3 | 1 | 0
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

26. Primary Outcome: Number of Teeth With Any Root Lesion From Radiography in 3 Groups
Description: Radiographic evaluation for any periapical or bifurcal lesion, cyst formation or obliteration
Time Frame: Change from Baseline at 3 months in 3 groups
Population: 1 tooth is extracted in HA group so 1 tooth is reduced but not participant
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth | 7 | 3 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

27. Primary Outcome: Number of Teeth With Any Root Lesion From Radiography in 3 Groups
Description: Radiographic evaluation for any periapical or bifurcal lesion, cyst formation or obliteration
Time Frame: Change from Baseline at 6 months in 3 groups
Population: 1 tooth exfoliated in FS group so 1 tooth and 1 participant are not evaluated in FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth | 4 | 4 | 3
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

28. Primary Outcome: Number of Teeth With Any Root Lesion From Radiography in 3 Groups
Description: Radiographic evaluation for any periapical or bifurcal lesion, cyst formation or obliteration
Time Frame: Change from Baseline at 12 months in 3 groups
Population: as for outcome 24
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 28 | 26 | 26
Number analyzed (teeth) | 35 | 32 | 31
teeth | 4 | 4 | 2
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

29. Secondary Outcome: Restoration Stability
Description: The survival rate of stainless steel crown and composite applied to each pulpotomized tooth
Time Frame: Change from Baseline at 1 month
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 51 | 40 | 39
teeth
  Stainless steel crown | 33 | 28 | 28
  Composite | 18 | 12 | 11
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

30. Secondary Outcome: Restoration Stability
Description: The survival rate of stainless steel crown and composite applied to each pulpotomized tooth
Time Frame: Change from Baseline at 3 months
Population: 1 tooth extracted from HA group so reduced to 50 teeth but no participant reduction
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 34
Number analyzed (teeth) | 50 | 40 | 39
teeth
  Stainless steel crown | 32 | 28 | 28
  Composite | 18 | 12 | 11
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

31. Secondary Outcome: Restoration Stability
Description: The survival rate of stainless steel crown and composite applied to each pulpotomized tooth
Time Frame: Change from Baseline at 6 months
Population: 1 tooth exfoliated from FS group so 1 tooth and 1 participant reduced from FS group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 50 | 40 | 38
teeth
  Stainless steel crown | 32 | 28 | 27
  Composite | 18 | 12 | 11
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

32. Secondary Outcome: Restoration Stability
Description: The survival rate of stainless steel crown and composite applied to each pulpotomized tooth
Time Frame: Change from Baseline at 12 months
Population: 2 teeth exfoliated from HA group so 50 teeth reduced to 48 teeth in HA group
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
Number analyzed (Participants) | 34 | 33 | 33
Number analyzed (teeth) | 48 | 40 | 38
teeth
  Stainless steel crown | 31 | 28 | 27
  Composite | 17 | 12 | 11
Statistical Analysis 1: Comparison: Hyaluronic Acid vs Formocresol vs Ferric Sulfate; Chi-Square Test was used to compare qualitative data.The results were evaluated at the significance level of p<0,05; Test type: Superiority; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Overall study;1st month,3rd month,6th month and 12th month after the treatments
Description: 1. pain or discomfort may be seen after the treatment of the primary tooth
  2. tooth can be exfoliated prematurely
Arm/Group | Hyaluronic Acid | Formocresol | Ferric Sulfate
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronic Acid (N=34) | Formocresol (N=33) | Ferric Sulfate (N=34)
pulpitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) — root canals of the primary molars can be inflamed and infected so that the patient can feel the pain or discomfort during chewing.

LIMITATIONS AND CAVEATS:
The limitations of this study included the unfortunate Covid-19 pandemic that interfered with the radiographic results of our study at 12th month, 8 participants did not show up to the dental appointments at 12th month and complicated the follow-up results on radiographs. However we managed to do the clinical examinations of all patients via social video conferencing devices (teledentistry).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04115358/Prot_SAP_000.pdf